CLINICAL TRIAL: NCT06888024
Title: Pelvic Vein Quantitative Flow Characterization Using 2D and 4D Flow MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningcheng Peter Li (Other)
Responsible Party: Sponsor-Investigator, Ningcheng Peter Li, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002051
Record Dates: First submitted 2025-02-12; First posted 2025-03-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: May-Thurner Syndrome; Iliac Venous Compression
Keywords: May-Thurner Syndrome; Iliac Venous Disease
MeSH Terms: conditions — May-Thurner Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with no imaging evidence of iliac venous disease (Experimental): Healthy volunteers with no self-reported history or prior imaging evidence of pelvic venous disease or associated symptoms to undergo 2D and 4D flow MRI without contrast administration
  Interventions: Procedure: non-contrast enhanced abdomen and pelvis MRI
- Patients with left iliac vein compression syndrome (a.k.a. May-Thurner syndrome). (Experimental): Patients with prior imaging evidence of left common iliac vein compression syndrome to undergo 2D and 4D flow MRI without contrast administration
  Interventions: Procedure: non-contrast enhanced abdomen and pelvis MRI
- Patients status post iliac stent placement (Experimental): Patients with a history of iliac stent placement to undergo 2D and 4D flow MRI without contrast administration
  Interventions: Procedure: non-contrast enhanced abdomen and pelvis MRI

INTERVENTIONS:
Procedure: non-contrast enhanced abdomen and pelvis MRI — non-contrast enhanced abdomen and pelvis MRI

SUMMARY:
The purpose of the study is to quantitatively characterize the flow in the pelvic venous structures using 2D and 4D flow MRI with the objective of establishing physiologic and pathologic parameters for downstream computational fluid dynamics analysis.

Arm 1: To establish the baseline flow characteristics of the iliac veins in patients with no imaging evidence of iliac venous disease.

Arm 2: To assess the flow characteristics of the iliac veins in patients with left iliac vein compression syndrome (a.k.a. May-Thurner syndrome).

Arm 3: To assess the flow characteristics of the iliac veins in patients status post iliac stent placement.

ELIGIBILITY:
Arm 1: Inclusion Criteria:

• No self-reported history of pelvic or iliac venous disease or associated symptoms

Exclusion Criteria:

* History of pelvic or iliac venous disease or intervention
* Contraindication to MRI examination
* Prisoners
* Subjects ≤ 18 years of age
* Pregnant women
* Adults unable to provide informed consent

Arm 2: Inclusion Criteria:

• Clinical symptoms or imaging findings compatible with left iliac vein compression syndrome

Exclusion Criteria:

* History of pelvic or iliac venous intervention
* Contraindication to MRI examination
* Prisoners
* Subjects ≤ 18 years of age
* Pregnant women
* Adults unable to provide informed consent

Arm 3: Inclusion Criteria:

• History of left iliac vein stent placement

Exclusion Criteria:

* Contraindication to MRI examination
* Prisoners
* Subjects ≤ 18 years of age
* Pregnant women
* Adults unable to provide informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Flow Volume | At Enrollment
  Flow volume in the iliac veins calculated based on the 2D and 4D flow MRI obtained.
12-month primary patency rate | 12 Months
  Freedom from occlusion of the stented segment; Freedom from restenosis >=50%; and Freedom from clinically-driven target lesion revascularization

SECONDARY OUTCOMES:
Flow Velocity Profile | At Enrollment
  Flow velocity profile in the iliac veins calculated based on the 2D and 4D flow MRI obtained.
Quality-of-life measure: Venous clinical severity score (VCSS) | Baseline to 6 Months, 12 Months, 24 Months, 36 Months
  Venous clinical severity scale (VCSS) is used to assess chronic venous disease (CVD) severity through clinical symptoms and signs. Ten areas are scored on a range from 0 (none) to 3 (severe), depending on the presence and severity of symptoms, signs, and the use of compression therapy. The scores for each of the ten items are then combined to calculate the total VCSS score with a higher score indicating more severe disease.
Quality-of-life measures | Baseline to 6 Months, 12 Months, 24 Months, 36 Months
  Chronic venous quality-of-life questionnaire (CIVIQ-20 Global Index)
Technical success | Index Procedure
  Successful delivery and deployment of the stent and removal of the delivery system during the index procedure
Target vessel revascularization | 30 days, 6 months, 12 months, 24 months, 36 months
  Determination of target vessel revascularization
Target lesion revascularization | 30 days, 6 months, 12 months, 24 months, 36 months
  Determination of target lesion revascularization
Major adverse events | 6 Months, 12 Months, 24 Months, 36 Months
  Identification of any major adverse events experienced
Clinical-etiologic-anatomic-pathophysiologic clinical score (CEAP) | Baseline to 6 Months, 12 Months, 24 Months, 36 Months
  CEAP score assessment
Primary Patency | 24 Months, 36 Months
  Freedom from occlusion of the stented segment of the target lesion; Freedom from restenosis ≥50% of the stented segment of the target lesion; Freedom from clinically driven target lesion revascularization.
Stent integrity | 30 Days, 12 Months, 24 Months, 36 Months
  Determination of integrity of the stent via scheduled visit-based evaluable imaging and unscheduled imaging

CONTACTS AND LOCATIONS:
Overall Officials: Ningcheng Li, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States